CLINICAL TRIAL: NCT00847054
Title: A Study of the Safety, Tolerability, and Pharmacokinetics of MORAb-004, a Humanized Monoclonal Antibody, in Subjects With Solid Tumors
Brief Title: A Study of of MORAb-004 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-004-001
Record Dates: First submitted 2009-02-05; First posted 2009-02-19 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Endosialin
MeSH Terms: interventions — ontuxizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MORAb-004 (Experimental)
  Interventions: Drug: MORAb-004 (monoclonal antibody to TEM1)

INTERVENTIONS:
Drug: MORAb-004 (monoclonal antibody to TEM1) — Intravenous administration

SUMMARY:
The purpose of this study is to determine the safety of multiple intravenous infusions of MORAb-004.

DETAILED DESCRIPTION:
MORAb-004 is a monoclonal antibody directed against endosialin, a cell surface glycoprotein, which is expressed on cells involved in tumor vasculature. Studies have found endosialin to play a key role in tumor growth and neovessel formation in numerous cancer types including (but not limited to) renal, breast, colon, pancreatic, lung, endometrial, ovarian, melanoma, sarcoma, and neuroectodermal tumors. Preclinical pharmacological studies have shown that MORAb-004 is a potentially useful anti-cancer agent. This clinical trial is being performed to determine the safety of MORAb-004 in subjects with solid tumors, as well as to establish serum pharmacokinetics of the antibody, and to assess tumor antigens that may serve as predictors of a response to MORAb-004. Study Part 2 was added to enroll subjects with specific histological diagnoses (colorectal cancer and soft tissue sarcoma) to further characterize the safety and tolerability of 5 dose levels of MORAb-004 previously tested during the dose escalation in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age.
* Subjects with any malignant solid tumor without intracranial involvement or metastases diagnosed by standard pathology criteria that has failed standard chemotherapy.
* Subject must have disease, as defined by RECIST or evaluable by clinical signs/symptoms (e.g., ascites, pleural effusion, or lesions of less than 2 cm) supported by biomarker, radiologic, or pathologic studies conducted within 4 weeks prior to study entry.
* Karnofsky performance status ≥70%.
* Female subjects of childbearing potential and all male subjects must consent to use a medically acceptable method of contraception throughout the study period and for 30 days after MORAb-004 administration. A barrier method of contraception must be included.
* Laboratory and clinical results within the 2 weeks prior to Study Day 1 as follows: Absolute neutrophil count (ANC) ≥1.5 x 109/L; Platelet count ≥100 x 109/L; Hemoglobin ≥10 g/dL; Serum bilirubin ≤2.0 mg/dL; Aspartate transaminase (AST) ≤2.5 x ULN; or ≤5 x ULN if liver metastases are present; Alanine transaminase (ALT) ≤2.5 x ULN; or ≤5 x ULN if liver metastases are present; Serum creatinine ≤2.0 mg/dL; prothrombin time (PT) and aPTT within institutional limits of normal.
* Subject must be willing and able to provide written informed consent.
* In Part 2 (expansion cohorts) ONLY, subjects must have a histological diagnosis of either CRC or STS (and subtypes, excluding bone sarcomas).

Exclusion Criteria:

* Known central nervous system (CNS) tumor involvement or metastases.
* Evidence of other active malignancy.
* Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class III or IV, angina not well controlled by medication, or myocardial infarction within 6 months).
* Electrocardiogram (ECG) demonstrating clinically significant arrhythmias (Note: Subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal SVT, are eligible).
* Presence of severe lung disease (In the absence of clinically apparent severe lung disease, no formal testing is necessary. In the presence of clinically severe lung disease, FEV1 must be >60% in order for the subject to be eligible.)
* Active serious systemic disease, including active bacterial or fungal infection.
* Chronic inflammatory disorder, e.g., inflammatory bowel disease, active vasculitis.
* Chemotherapy, biologic therapy, or immunotherapy within 3 weeks prior to enrollment.
* Breast-feeding, pregnant, or likely to become pregnant during the study.
* Active hepatitis or human immunodeficiency virus (HIV) infection.
* Subjects who have received a previous monoclonal antibody therapy and have evidence of an immune or allergic reaction, or previously documented human anti-human antibody (HAHA).
* Subjects with large ascites or pleural effusion (≥500 cc) based on results of most recent CT scan).
* Chronic systemic anticoagulation therapy with warfarin or heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety of multiple intravenous infusions of MORAb-004 | Weekly while receiving study drug
  Safety is evaluated by clinical assessment, monitoring of adverse events, laboratory evaluations, ECG.

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of MORAb-004 (within the administered range) | Weekly
  Monitoring of adverse events, laboratory test results and ECG results.
To determine optimal biologic dose (OBD) of MORAb-004 | Weekly
  Monitoring of adverse events, laboratory evaulations and ECG results.
To establish the serum pharmacokinetics of MORAb-004 using a validated assay | Weekly
  Serial serum PK evaluations.
To describe changes in the objective measurements of tumor size and biomarkers (if applicable)after treatment with MORAb-004 | bimonthly
  CT or MRI evaluations following every other 4-week cycle.
To detect any antibody response (human anti-human antibodies [HAHA] to multiple intravenous infusions of MORAb-004 | Biweekly
  Biweekly serum collection for detection of HAHA during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Weil, MD, Study Director — Morphotek
Locations (3):
- United States (3):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania